CLINICAL TRIAL: NCT03405402
Title: Transfusion in Sickle Cell Disease: Risk Factors for Alloimmunization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanane EL KENZ (Other)
Responsible Party: Sponsor-Investigator, Hanane EL KENZ, Head of Blood Bank, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CHUB-PRO-TRANSFU-DREPANO 1
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease; Allo-immunization; Blood transfusion
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Allo-immunization detected (positive response for irregular antibodies 2 to 4 weeks after a blood transfusion)
  Interventions: Procedure: Blood sampling
- Control group (Other): Allo-immunization not detected
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Extra blood sampling at the time of a blood transfusion in order to perform the laboratory analysis

SUMMARY:
Sickle cell patients have a high prevalence of alloimmunization. This high rate of alloimmunization can be partially explained by the existence of an antigenic difference between the predominantly Caucasian donor population and the sickle cell patients of African origin. Genetic and environmental risk factors have also been described.

The main risk factors that have been shown in retrospective or cross-sectional studies are some HLA alleles, the age of the patient, the number of leukocyte-depleted erythrocyte concentrates (CED) transfused, the number of transfusion episodes, the age of the CEDs, the existence of an inflammatory event at the time of transfusion and the presence of anti-erythrocyte autoantibodies.There is also evidence of an impaired TH response but the underlying immunological mechanism is not fully understood.

The aim of this study is to study the prevalence and the risk factors for anti-erythrocyte alloimmunization and to try to understand the immunological mechanisms.

ELIGIBILITY:
Inclusion Criteria:

Sickle cell disease patients treated within the CHU Brugmann or Queen Fabiola Children's Hospital

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
Irregular antibodies | 1 hour before blood transfusion
  Presence/abscence of irregular antibodies
Irregular antibodies | Between 2 to 4 weeks after blood transfusion
  Presence/abscence of irregular antibodies
C-reactive protein (CRP) | 1 hour before blood transfusion
  CRP dosage
Cytokine | 1 hour before blood transfusion
  Cytokine dosage
Cytokine | Between 2 to 4 weeks after blood transfusion
  Cytokine dosage
Heme oxygenase | 1 hour before blood transfusion
  Heme oxygenase dosage
Heme oxygenase | Between 2 to 4 weeks after blood transfusion
  Heme oxygenase dosage
Lymphocyte typing | 1 hour before blood transfusion
  Lymphocyte typing
Lymphocyte typing | Between 2 to 4 weeks after blood transfusion
  Lymphocyte typing

SECONDARY OUTCOMES:
Sex | 1 hour before blood transfusion
  Sex
Chronic or acute blood transfusion | 1 hour before blood transfusion
  Blood transfusions planned at regular intervals of time (chronic transfusions) or performed in reaction to a medical issue (acute transfusion).
Blood transfusion indication | 1 hour before blood transfusion
  Medical reason explaining the necessity of a blood transfusion
Blood donor ethnicity | 1 hour before blood transfusion
  Blood donor ethnicity

CONTACTS AND LOCATIONS:
Overall Officials: Marie Deleers, Ph Biol, Principal Investigator — CHU Brugmann
Locations (2):
- Belgium (2):
  - CHU Brugmann, Brussels
  - HUDERF, Brussels

IPD SHARING:
Plan to Share IPD: No